CLINICAL TRIAL: NCT05284578
Title: The Effects of Expressive Writing and Compassionate Letter Writing on Emotional Distress Intolerance: A Brief Randomized Controlled Trial
Brief Title: The Effects of Expressive Writing and Compassionate Letter Writing on Emotional Distress Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Allison Kelly, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42863
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Distress Intolerance

STUDY DESIGN:
Intervention Model Description: 1/3 of the study participants (43 from UWaterloo, 98 from Prolific) were placed into the self-compassionate writing intervention group, 1/3 of the study participants (42 from UWaterloo, 100 from Prolific) were placed into the expressive writing intervention group, and 1/3 of the study participants (41 from UWaterloo, 100 from Prolific) were placed into the control group.
Who Masked: Participant
Masking Description: The participant did not know prior to their study participation that there are three different study conditions, and they did not find out which condition they were randomized to until the end of their study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-compassionate writing intervention (Experimental): Participants assigned to this intervention were asked to engage in one brief online self-compassionate writing session, where they were asked to write about and experience their feelings from the perspective of an inner compassionate observer.
  Interventions: Other: Self-compassionate writing intervention
- Expressive writing intervention (Experimental): Participants assigned to this intervention were asked to engage in one brief online expressive writing session, where they were asked to explore their deepest thoughts and emotions surrounding an upsetting situation through writing.
  Interventions: Other: Expressive writing intervention
- Control writing task (Active Comparator): Participants assigned to this condition were asked to engage in a neutral time management writing task.
  Interventions: Other: Control writing task

INTERVENTIONS:
Other: Self-compassionate writing intervention — Participants assigned to this intervention were asked to engage in one brief online self-compassionate writing session, where they were asked to write about and experience their feelings from the perspective of an inner compassionate observer.
  Arms: Self-compassionate writing intervention
Other: Expressive writing intervention — Participants assigned to this intervention were asked to engage in one brief online expressive writing session, where they were asked to explore their deepest thoughts and emotions surrounding an upsetting situation through writing.
  Arms: Expressive writing intervention
Other: Control writing task — Participants assigned to this condition were asked to engage in a neutral time management writing task.
  Arms: Control writing task

SUMMARY:
Perceived emotional distress intolerance is a transdiagnostic marker of psychopathology associated with psychological and interpersonal dysfunction, and the development of interventions for perceived emotional distress intolerance is of prime importance. One potential intervention is a behavioural experiment, i.e. a cognitive behaviour therapy technique where clients undergo an exercise designed to test a maladaptive belief, e.g., that negative emotions are unbearable, and adjust their belief to accommodate any disconfirmatory information that arises through the exercise. This study examines the effects of a one-session self-compassion writing behavioural experiment compared to a one-session expressive writing behavioural experiment on low perceived distress tolerance. Participants were recruited from the University of Waterloo and Prolific, and were randomly assigned to the self-compassion condition, expressive writing condition, or a control condition.

DETAILED DESCRIPTION:
The study consisted of two online surveys. During the first survey, participants answered a set of questionnaires. Then, they were prompted to think of an upsetting situation and the associated unpleasant emotions, and they were then randomly assigned to a brief self-compassionate writing, expressive writing, or neutral writing task. They then answered a series of questionnaires immediately after completing the writing task. During the second survey, one week later, participants answered a brief set of questionnaires.

ELIGIBILITY:
Inclusion Criteria for University of Waterloo sample:

* Undergraduate students with a SONA account who are high in emotional distress intolerance (i.e. a lower-than-average score on the Distress Tolerance Scale; mean based on SONA student sample)

Inclusion Criteria for Prolific sample:

* Adults with a Prolific account who are high in emotional distress intolerance (i.e. a lower-than-average score on the Distress Tolerance Scale; mean based on Prolific sample)
* First language English speakers

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Distress Tolerance Scale | Change from baseline to one week post-intervention
  Self-report questionnaire with 15 questions on a 5-point Likert scale (scored 1-5, with 4 subscales). Mean scores range from 1-5, with higher increase in score indicative of increased perceived distress tolerance.
Distress Tolerance Scale (short form) | Immediately post-intervention
  Self-report questionnaire with 4 questions on a 5-point Likert scale (scored 1-5). Mean scores range from 1-5, with higher score indicative of greater perceived distress tolerance.
Endorsement and Discomfort Scale (adapted) | Immediately post-intervention
  Self-report questionnaire with 10 questions on a 9-point Likert scale (scored 1-9). Total scores range from 10-90, with higher score indicative of greater acceptability of intervention.
Endorsement and Discomfort Scale (adapted) | One week post-intervention
  Self-report questionnaire with 10 questions on a 9-point Likert scale (scored 1-9). Total scores range from 10-90, with higher score indicative of greater acceptability of intervention.
Compassionate Engagement and Action Scale | Change from baseline to one week post-intervention
  Self-report questionnaire with 13 questions on a 10-point Likert scale (scored 1-10). Three questions are reverse-scored and not included in scoring. Total scores range from 10-100, with higher increase in score indicative of increased emotional engagement

SECONDARY OUTCOMES:
Soothing affect measures (researcher-generated) - Adapted from the Serenity Subscale of the PANAS-X and the Safe/Warmth Positive Affect Subscale of the Types of Positive Affect Scale (TPAS) | Immediately post-intervention (assessed as a mediator)
  Self-report questionnaire with 7 questions on a 5-point Likert scale (scored 1-5). Total scores range from 7-35, with higher score indicative of more soothing affect.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kelly, PhD, Principal Investigator — Associate professor
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada